CLINICAL TRIAL: NCT00474253
Title: A Multicenter, Randomized, Parallel Group, Comparative, Active-Controlled, Safety-Assessor Blinded, Phase IIIa, Trial, in Adult Subjects Comparing Recovery From 1.2 mg.Kg-1 Rocuronium Followed by 16 mg.Kg-1 Org 25969 at 3 Minutes With Recovery From 1.0 mg.Kg-1 Succinylcholine
Brief Title: Comparison of Recovery From Rocuronium 1.2 mg/kg Followed by Sugammadex (Org 25969) 16 mg/kg at 3 Minutes With Recovery From Succinylcholine 1.0 mg/kg (19.4.303)(P05946)(MK-8616-026)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05946; 19.4.303 (Other: Organon Protocol Number); P05946 (Other: Schering-Plough Protocol Number); MK-8616-026 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Succinylcholine; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rocuronium + Sugammadex (Experimental): Participants were to receive a single bolus dose of 1.2 mg/kg rocuronium. Three minutes after the start of the rocuronium administration, they were to receive a single bolus dose of 16.0 mg/kg sugammadex.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Succinylcholine (Active Comparator): Participants were to receive a single bolus dose of 1.0 mg/kg succinylcholine and allowed to recovery spontaneously from neuromuscular blockade.
  Interventions: Drug: Succinylcholine

INTERVENTIONS:
Drug: Sugammadex — Single bolus intravenous (IV) dose of 16.0 mg/kg sugammadex
  Other Names: Org 25969; MK-8616
  Arms: Rocuronium + Sugammadex
Drug: Succinylcholine — Single bolus IV dose of 1.0 mg/kg succinylcholine
  Arms: Succinylcholine
Drug: Rocuronium — Single bolus IV dose of 1.2 mg/kg rocuronium
  Other Names: Zemuron®
  Arms: Rocuronium + Sugammadex

SUMMARY:
The purpose of the trial is to demonstrate a faster recovery from neuromuscular block induced by 1.2 mg/kg rocuronium after reversal at 3 minutes by 16.0 mg/kg of sugammadex compared with recovery after a neuromuscular block induced by 1.0 mg/kg succinylcholine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 or 2 physical status;
* 18 to 65 years of age (inclusive);
* Scheduled for elective surgical procedure under general anesthesia requiring a short duration of neuromuscular block with the use of rocuronium or succinylcholine and requiring endotracheal intubation;
* Scheduled for surgery in supine position;
* Body mass index (BMI) < 30;
* Given written informed consent.

Exclusion Criteria:

* Has ischemic heart disease or history of myocardial infarction within the last year;
* May experience difficult intubation due to anatomical malformations;
* Known or suspected to have neuromuscular disorders impairing neuromuscular blockade and/or significant renal dysfunction;
* Known or suspected family history of malignant hyperthermia;
* Known or suspected allergy to narcotics, muscle relaxants, midazolam, anesthetics or other medications used during surgery;
* Is receiving medication known to interfere with neuromuscular blocking agents such as anticonvulsants, antibiotics and Mg2+;
* Individuals in whom the use of neostigmine and/or glycopyrrolate may be contraindicated;
* Females who are pregnant or breast-feeding;
* Females of childbearing potential who are not using an acceptable method of birth control [condom or diaphragm with spermicide, vasectomized partner (> 6 months), IUD, abstinence];
* Has already participated in a sugammadex trial including Protocol 19.4.303.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-02-10 (Actual); Primary Completion 2006-08-22 (Actual); Study Completion 2006-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Lee C, Jahr JS, Candiotti KA, Warriner B, Zornow MH, Naguib M. Reversal of profound neuromuscular block by sugammadex administered three minutes after rocuronium: a comparison with spontaneous recovery from succinylcholine. Anesthesiology. 2009 May;110(5):1020-5. doi: 10.1097/ALN.0b013e31819dabb0. PMID 19387176
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Rocuronium + Sugammadex: Participants received a single bolus intravenous (IV) dose of 1.2 mg/kg rocuronium to induce neuromuscular block. This was followed by a single bolus IV dose of sugammadex 16.0 mg/kg three minutes after the start of rocuronium administration, to reverse the neuromuscular block.
- Succinylcholine: Participants received a single bolus IV dose of 1.0 mg/kg succinylcholine to induce neuromuscular block. They were allowed to recovery spontaneously from the neuromuscular block.
Period: Overall Study
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Started | 58 (Includes 2 participants randomized to succinylcholine group who received rocuronium + sugammadex.) | 57 (Includes 1 participant randomized to rocuronium + sugammadex group who received succinylcholine.)
Treated | 56 (Based on actual treatment received.) | 54 (Based on actual treatment received.)
Completed | 55 (Based on actual treatment received.) | 53 (Based on actual treatment received.)
Not Completed | 3 | 4
Not completed — Withdrew consent | 2 | 0
Not completed — Withdrew due to surgery-related issues | 0 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discharged prior to study completion | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received study treatment
Groups:
- Rocuronium + Sugammadex: Participants received a single bolus IV dose of 1.2 mg/kg rocuronium to induce neuromuscular block. This was followed by a single bolus IV dose of sugammadex 16.0 mg/kg 3 minutes after the start of rocuronium administration, to reverse the neuromuscular block.
- Total: Total of all reporting groups
Arm/Group | Rocuronium + Sugammadex | Succinylcholine | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (13) | 41 (13) | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery of T1 to 10% of Baseline Value From Start of Rocuronium + Sugammadex or Succinylcholine Administration
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 refers to the amplitude (height) of the first twitch after TOF nerve stimulation.
Time Frame: Up to 15 minutes after administration of rocuronium + sugammadex or succinylcholine
Population: All participants who received study treatment and had at least one post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 54 | 53
Minutes | 4.35 (0.72) | 7.15 (1.55)

2. Secondary Outcome: Time to Recovery of T1 to 90% of Baseline Value From Start of Rocuronium + Sugammadex or Succinylcholine Administration
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 refers to the amplitude (height) of the first twitch after TOF nerve stimulation.
Time Frame: Up to 20 minutes after administration of rocuronium + sugammadex or succinylcholine
Population: All participants who received study treatment and had at least one post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 54 | 53
Minutes | 6.13 (1.78) | 11.03 (2.40)

3. Secondary Outcome: Level of Consciousness: Number of Participants Awake and Oriented
Description: The number of participants who were awake and oriented was assessed as part of an overall assessment of the clinical level of consciousness. The clinical level of consciousness was used as a measure of recovery from neuromuscular blockade at two time points: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. Attempts were made to arouse participants every 15 minutes with mild prodding, mild shaking, and asking questions regarding name, location, and day of the week. The assessment ended once the participant was awake and fully orientated.
Time Frame: Up to 24 hours after administration of rocuronium + sugammadex or succinylcholine
Population: All participants who received study treatment, had at least one post-baseline efficacy measurement, and had no major protocol violations
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 32 | 41
Participants
  Prior to transfer to recovery room | 8 | 13
  Prior to discharge from recovery room | 19 | 33

4. Secondary Outcome: Level of Consciousness: Number of Participants Arousable With Minimal Stimulation
Description: The number of participants aroused with minimal stimulation was assessed as part of an overall assessment of level of consciousness. The level of consciousness was used as a measure of recovery from neuromuscular blockade at two time points: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. Attempts were made to arouse participants every 15 minutes with mild prodding, mild shaking, and asking questions regarding name, location, and day of the week. The assessment ended once the participant was awake and fully orientated.
Time Frame: Up to 24 hours after administration of rocuronium + sugammadex or succinylcholine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 32 | 41
Participants
  Prior to transfer to recovery room | 7 | 15
  Prior to discharge from recovery room | 1 | 2

5. Secondary Outcome: Level of Consciousness: Number of Participants Responsive Only to Tactile Stimulation
Description: The number of participants responsive only to tactile stimulation was assessed as part of an overall assessment of the level of consciousness. The level of consciousness was used as a measure of recovery from neuromuscular blockade at two time points: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. Attempts were made to arouse participants every 15 minutes with mild prodding, mild shaking, and asking questions regarding name, location, and day of the week. The assessment ended once the participant was awake and fully orientated.
Time Frame: Up to 24 hours after administration of rocuronium + sugammadex or succinylcholine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 32 | 41
Participants
  Prior to transfer to recovery room | 5 | 7
  Prior to discharge from recovery room | 0 | 0

6. Secondary Outcome: Number of Participants Able to Perform 5-Second Head Lift
Description: The number of participants who were able to lift their head for 5 seconds was assessed as a measure of recovery following neuromuscular blockade at two time points: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. The assessment was performed every 15 minutes until the first successful 5-second head lift was achieved.
Time Frame: Up to 24 hours after administration of rocuronium + sugammadex or succinylcholine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 32 | 41
Participants
  Prior to transfer to recovery room | 13 | 24
  Prior to discharge from recovery room | 20 | 35

7. Secondary Outcome: Number of Participants Experiencing General Muscle Weakness
Description: The number of participants experiencing general muscle weakness was assessed by the investigator as a measure of recovery from neuromuscular blockade at two time points: prior to transfer to the recovery room after extubation and prior to discharge from the recovery room. The assessments were performed every 15 minutes until the absence of general muscle weakness. A standardized examination form was used to determine the presence or absence of muscle weakness in various muscle groups.
Time Frame: Up to 24 hours after administration of rocuronium + sugammadex or succinylcholine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
Number analyzed (Participants) | 32 | 41
Participants
  Prior to transfer to recovery room | 2 | 3
  Prior to discharge from recovery room | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 days after administration of rocuronium + sugammadex or succinylcholine
Description: All participants who received study treatment
Arm/Group | Rocuronium + Sugammadex | Succinylcholine
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/54
Other Adverse Events (participants affected / at risk) | 51/56 | 50/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex (N=56) | Succinylcholine (N=54)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex (N=56) | Succinylcholine (N=54)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 16 (20) | 20 (23)
Vomiting (Gastrointestinal disorders) | 9 (9) | 8 (8)
Chills (General disorders) | 6 (6) | 7 (7)
Pyrexia (General disorders) | 5 (6) | 5 (8)
Incision site complication (Injury, poisoning and procedural complications) | 5 (5) | 7 (10)
Procedural complication (Injury, poisoning and procedural complications) | 5 (7) | 4 (4)
Procedural hypertension (Injury, poisoning and procedural complications) | 7 (8) | 7 (7)
Procedural hypotension (Injury, poisoning and procedural complications) | 7 (7) | 13 (14)
Procedural pain (Injury, poisoning and procedural complications) | 32 (34) | 26 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (9)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 8 (9) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (4)
Urinary retention (Renal and urinary disorders) | 2 (2) | 4 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning this clinical trial will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.